CLINICAL TRIAL: NCT03338010
Title: A Prospective, Randomized, Open-Label Comparison of a Long-Acting Basal Insulin Analog LY2963016 to Lantus® in Adult Chinese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2963016 Compared to Lantus® in Adult Chinese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16037; I4L-GH-ABET (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes
Keywords: Insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY2963016 (Experimental): Insulin naive participants started on 10 units (U) LY2963016 given subcutaneously (SC) once a day (QD) for 24 weeks. Participants-driven titration was supervised by investigators through the course of the study to maintain the fasting blood glucose (FBG) ≤100 milligram per deciliter (mg/dL) (5.6 millimoles per litre [mmol/L]) while avoiding hypoglycemia. Participants were allowed to continue oral antihyperglycemic medication (OAM).
  Interventions: Drug: LY2963016
- Lantus® (Active Comparator): Insulin naive participants started on 10 U Lantus® given SC QD for 24 weeks. Participants-driven titration was supervised by investigators through the course of the study to maintain the FBG ≤100 mg/dL (5.6 mmol/L) while avoiding hypoglycemia. Participants were allowed to continue oral OAM.
  Interventions: Drug: Lantus®

INTERVENTIONS:
Drug: LY2963016 — Administered SC
  Arms: LY2963016
Drug: Lantus® — Administered SC
  Arms: Lantus®

SUMMARY:
The purpose of this study is to compare long-acting basal insulin analog LY2963016 to Lantus® in insulin naïve adult Chinese participants with Type 2 Diabetes Mellitus (T2DM) on 2 or more oral antihyperglycemic medications (OAMs). Participants will continue their OAMs throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM based on the disease diagnostic criteria World Health Organization (WHO) classification.
* Have been receiving 2 or more OAMs at stable doses for the 12 weeks prior to screening.
* Have a HbA1c ≥7.0% and ≤11.0%.
* Body mass index (BMI) ≤35 kilograms per meter squared.

Exclusion Criteria:

* Have used insulin therapy (outside of pregnancy) anytime in the past 1 year, except for short-term treatment of acute conditions, and up to a maximum of 4 continuous weeks.
* Have used any glucagon like peptide (GLP-1) receptor agonists within the previous 90 days.
* Are currently taking traditional medicine (herbal medicine or patent medicine) with known/specified content of anti-hyperglycemic effects within 3 months before screening.
* Have had more than one episode of severe hypoglycemia within 6 months prior to entry into the study.
* Have had ≥2 emergency room visits or hospitalizations due to poor glucose control.
* Have known hypersensitivity or allergy to Lantus® or its excipients.
* Are receiving chronic systemic glucocorticoid therapy at pharmacological doses or have received such therapy within 4 weeks immediately preceding screening.
* Have obvious signs or symptoms, or laboratory evidence, of liver disease.
* Have one of the following concomitant diseases: significant cardiac or gastrointestinal disease.
* Have a history of renal transplantation, are currently receiving renal dialysis or have a serum creatinine greater than 2.0 milligrams per deciliter.
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia.
* Participants with active cancer or personal history of cancer within the previous 5 years.
* Are pregnant or intend to become pregnant during the course of the study.
* Are women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- China (32):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun-Yat Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shantou University Medical College No.2 Affiliated Hospital, Shantou, Guangdong
  - The 1st Affiliated Hospital of Henan Science and technology, Luoyang, Henan
  - Wuhan Central Hospital, Wuhan, Hubei
  - Tongji Hosp Tongji Med Col Huazhong Univ of Sci & Tech, Wuhan, Hubei
  - The First People Hospital of Yueyang, Yueyang, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Affliated Jiangyin Hospital of Southeast University Medical College, Jiangyin, Jiangsu
  - Nanjing Drum Tower Hosp Affiliated Hosp of Nanjing Univ Med, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Xuzhou central Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Siping central people's hospital, Siping, Jilin
  - Dalian Med. Univ. No 2 Affiliate Hospital, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital with Nanjing Medical Universit, Nanjing, Nanjing
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Jinan Central Hospital, Jinan, Shandong
  - 1st affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Beijing
  - Chongqing General Hospital, Chongqing
  - Shanghai Putuo District Center Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2963016: Insulin naive participants started on 10 units (U) LY2963016 given subcutaneously (SC) once a day (QD) for 24 weeks. Participants-driven titration was supervised by investigators through the course of the study to maintain the fasting blood glucose (FBG) ≤ 100 milligram per deciliter (mg/dL) (5.6 millimoles per litre [mmol/L]) while avoiding hypoglycemia. Participants were allowed to continue oral antihyperglycemic medication (OAM).
Period: Overall Study
Arm/Group | LY2963016 | Lantus®
Started | 359 | 177
Received at Least One Dose of Study Drug | 359 | 177
Completed | 336 | 159
Not Completed | 23 | 18
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Lost to Follow-up | 4 | 2
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Non-Compliance with Study Drug | 0 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- LY2963016: Insulin naive participants started on 10 U LY2963016 given SC QD for 24 weeks. Participants-driven titration was supervised by investigators through the course of the study to maintain the FBG ≤100 mg/dL (5.6 mmol/L) while avoiding hypoglycemia. Participants were allowed to continue OAM.
- Total: Total of all reporting groups
Arm/Group | LY2963016 | Lantus® | Total
Number analyzed (Participants) | 359 | 177 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.6) | 59.5 (8.9) | 58.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 79 | 229
  Male | 209 | 98 | 307
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 359 | 177 | 536
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 359 | 177 | 536
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.42 (1.04) | 8.39 (0.92) | 8.41 (1.00)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 10.09 (5.47) | 10.69 (5.94) | 10.29 (5.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (LY2963016 to Lantus®)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least square (LS) mean was calculated by mixed-effects model for repeated measures (MMRM) with baseline, insulin secretagogues at study entry, treatment, visit and treatment*visit in the model.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least one non-missing post-baseline HbA1c value.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 334 | 158
Percentage of HbA1c | -1.27 (0.043) | -1.23 (0.062)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Non-Inferiority — 0.40% noninferiority margin was used; p = 0.545, Mixed Models Analysis; LS Mean Difference = -0.05, 95% CI 2-sided [-0.19 to 0.10]

2. Secondary Outcome: Change From Baseline in HbA1c (Lantus® to LY2963016)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean was calculated by MMRM with baseline, insulin secretagogues at study entry, treatment, visit and treatment*visit in the model.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 334 | 158
Percentage of HbA1c | -1.27 (0.043) | -1.23 (0.062)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Non-Inferiority — 0.40% noninferiority margin was used; p = 0.545, Mixed Models Analysis; LS Mean Difference = -0.05, 95% CI 2-sided [-0.19 to 0.10]

3. Secondary Outcome: Change From Baseline in 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: Seven-point SMBG are completed at the following timepoints: Before Morning Meal, 2 Hours After Morning Meal, Before Mid-Day Meal, 2 Hours After Mid-Day Meal, Before Evening Meal, 2 Hours After Evening Meal and Bed Time. LS mean was calculated by MMRM with baseline, insulin secretagogues at study entry, baseline HbA1c, treatment, time and treatment*time in the model.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and at least one non-missing post-baseline SMBG value.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 337 | 159
milligrams per deciliter (mg/dL)
  Before Morning Meal Glucose | -48.7 (1.09) | -49.7 (1.59)
  2 Hours After Morning Meal Glucose: number analyzed (Participants) | 328 | 155
  2 Hours After Morning Meal Glucose | -56.3 (2.34) | -52.7 (3.39)
  Before Mid-Day Meal Glucose: number analyzed (Participants) | 327 | 156
  Before Mid-Day Meal Glucose | -43.2 (2.03) | -39.9 (2.93)
  2 Hours After Mid-Day Meal Glucose: number analyzed (Participants) | 321 | 154
  2 Hours After Mid-Day Meal Glucose | -31.0 (2.31) | -35.9 (3.33)
  Before Evening Meal Glucose: number analyzed (Participants) | 325 | 155
  Before Evening Meal Glucose | -32.1 (2.21) | -33.0 (3.19)
  2 Hours After Evening Meal Glucose: number analyzed (Participants) | 320 | 153
  2 Hours After Evening Meal Glucose | -29.7 (2.46) | -32.0 (3.55)
  Bedtime Glucose: number analyzed (Participants) | 309 | 146
  Bedtime Glucose | -31.6 (2.35) | -33.0 (3.40)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Before Morning Meal Glucose; Test type: Superiority; p = 0.602, Mixed Models Analysis; LS Mean Difference = 1.0, 95% CI 2-sided [-2.8 to 4.8]
Statistical Analysis 2: Comparison: LY2963016 vs Lantus®; 2 Hours After Morning Meal Glucose; Test type: Superiority; p = 0.373, Mixed Models Analysis; LS Mean Difference = -3.7, 95% CI 2-sided [-11.8 to 4.4]
Statistical Analysis 3: Comparison: LY2963016 vs Lantus®; Before Mid-Day Meal Glucose; Test type: Superiority; p = 0.351, Mixed Models Analysis; LS Mean Difference = -3.3, 95% CI 2-sided [-10.3 to 3.7]
Statistical Analysis 4: Comparison: LY2963016 vs Lantus®; 2 Hours After Mid-Day Meal Glucose; Test type: Superiority; p = 0.230, Mixed Models Analysis; LS Mean Difference = 4.9, 95% CI 2-sided [-3.1 to 12.8]
Statistical Analysis 5: Comparison: LY2963016 vs Lantus®; Before Evening Meal Glucose; Test type: Superiority; p = 0.819, Mixed Models Analysis; LS Mean Difference = 0.9, 95% CI 2-sided [-6.7 to 8.5]
Statistical Analysis 6: Comparison: LY2963016 vs Lantus®; 2 Hours After Evening Meal Glucose; Test type: Superiority; p = 0.588, Mixed Models Analysis; LS Mean Difference = 2.3, 95% CI 2-sided [-6.2 to 10.9]
Statistical Analysis 7: Comparison: LY2963016 vs Lantus®; Bedtime Glucose; Test type: Superiority; p = 0.732, Mixed Models Analysis; LS Mean Difference = 1.4, 95% CI 2-sided [-6.7 to 9.5]

4. Secondary Outcome: Percentage of Participants With HbA1c <7% at Week 24
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 334 | 158
Percentage of participants | 43.7 | 44.9
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.846, Fisher Exact

5. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5% at Week 24
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 334 | 158
Percentage of participants | 23.4 | 16.5
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.098, Fisher Exact

6. Secondary Outcome: Change From Baseline in Glycemic Variability of Fasting Blood Glucose
Description: Glycemic variability is measured by the intra-participant standard deviation (SD) value of fasting blood glucose as measured by the actual morning and daily pre-meal blood glucose value from the 7-point self-monitoring blood glucose [SMBG] profiles. LS mean was calculated by MMRM with baseline, insulin secretagogues at study entry, baseline HbA1c, treatment, time and treatment*time in the model.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least one non-missing post-baseline SMBG value.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 327 | 157
milligrams per deciliter (mg/dL)
  Morning Pre-meal Standard Deviation: number analyzed (Participants) | 316 | 150
  Morning Pre-meal Standard Deviation | -2.17 (0.606) | -2.49 (0.879)
  Daily Mean Standard Deviation | -4.1 (0.85) | -4.5 (1.22)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Morning Pre-meal Standard Deviation; Test type: Superiority; p = 0.767, Mixed Models Analysis; LS Mean Difference = 0.32, 95% CI 2-sided [-1.78 to 2.42]
Statistical Analysis 2: Comparison: LY2963016 vs Lantus®; Daily Mean Standard Deviation; Test type: Superiority; p = 0.781, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-2.5 to 3.3]

7. Secondary Outcome: Basal Insulin Dose Units Per Day
Description: Units of basal insulin dose taken per day (U/day). LS mean was calculated by MMRM with baseline, insulin secretagogues at study entry, baseline HbA1c, treatment, time and treatment*time in the model.
Time Frame: At Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least one non-missing post-baseline basal Insulin dose value.
Measure: Least Squares Mean (Standard Error); unit: units per day (U/day)
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 341 | 161
units per day (U/day) | 16.0 (0.43) | 15.7 (0.61)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.750, Mixed Models Analysis; LS Mean Difference = 0.2, 95% CI 2-sided [-1.2 to 1.7]

8. Secondary Outcome: Change From Baseline in Basal Insulin Dose Units Per Day
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: U/day
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 341 | 161
U/day | 7.0 (0.43) | 6.8 (0.61)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.750, Mixed Models Analysis; LS Mean Difference = 0.2, 95% CI 2-sided [-1.2 to 1.7]

9. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was evaluated. LS mean was calculated by MMRM with baseline, insulin secretagogues at study entry, baseline HbA1c, treatment, time and treatment*time in the model.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and at least one non-missing post-baseline body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 334 | 158
kilogram (kg) | 1.1 (0.13) | 1.2 (0.19)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.3]

10. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ)
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. Items divided into 5 domains of satisfaction: Inconvenience of Regimen [(IR) 5 items: domain scores range (DSR) 5-35], Lifestyle Flexibility [(LF) 3 items: DSR 3-21], Glycemic Control [(GC) 3 items: DSR 3-21], Hypoglycemic Control [(HC) 5 items: DSR 5-35], Insulin Delivery Device [(IDD) 6 items: DSR 6-42]. All items measured on a 7-point scale: 1 (no bother at all) to 7 (a tremendous bother), with lower scores reflecting better outcomes. ITSQ Total Overall Raw Scores range from 22-154. Both raw domain and overall scores are transformed on a scale of 0-100, where transformed score=100*[(7-mean raw score)/6]. Higher scores indicate better treatment satisfaction. LS mean was calculated by MMRM with baseline, insulin secretagogues at study entry, baseline HbA1c, treatment, time and treatment*time in the model.
Time Frame: At Week 24
Population: All randomized participants who received at least 1 dose of study drug and had evaluable ITSQ data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 334 | 158
units on a scale
  IR | 89.36 (0.80) | 90.31 (1.16)
  LF | 83.70 (1.05) | 87.69 (1.52)
  HC | 89.07 (0.79) | 90.86 (1.15)
  GC | 87.80 (0.84) | 87.83 (1.21)
  IDD | 86.84 (0.86) | 88.29 (1.24)
  ITSQ Overall Total | 87.32 (0.75) | 88.99 (1.08)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Inconvenience of Regimen Transformed Score; Test type: Superiority; p = 0.500, Mixed Models Analysis; LS Mean Difference = -0.95, 95% CI 2-sided [-3.72 to 1.82]
Statistical Analysis 2: Comparison: LY2963016 vs Lantus®; Lifestyle Flexibility Transformed Score; Test type: Superiority; p = 0.031, Mixed Models Analysis; LS Mean Difference = -3.99, 95% CI 2-sided [-7.62 to -0.36]
Statistical Analysis 3: Comparison: LY2963016 vs Lantus®; Hypoglycemic Control Transformed Score; Test type: Superiority; p = 0.200, Mixed Models Analysis; LS Mean Difference = -1.79, 95% CI 2-sided [-4.53 to 0.95]
Statistical Analysis 4: Comparison: LY2963016 vs Lantus®; Glycemic Control Transformed Score; Test type: Superiority; p = 0.988, Mixed Models Analysis; LS Mean Difference = -0.02, 95% CI 2-sided [-2.92 to 2.88]
Statistical Analysis 5: Comparison: LY2963016 vs Lantus®; Insulin Delivery Device Satisfaction Transformed Score; Test type: Superiority; p = 0.337, Mixed Models Analysis; LS Mean Difference = -1.45, 95% CI 2-sided [-4.41 to 1.51]
Statistical Analysis 6: Comparison: LY2963016 vs Lantus®; ITSQ Overall Total; Test type: Superiority; p = 0.205, Mixed Models Analysis; LS Mean Difference = -1.67, 95% CI 2-sided [-4.26 to 0.92]

11. Secondary Outcome: Number of Participants With Detectable Anti-Glargine Antibodies
Description: Number of participants with detectable anti-glargine antibodies were reported.
Time Frame: Baseline through 24 weeks
Population: All randomized participants who received at least 1 dose of study drug. Only participants with detected insulin antibody levels at baseline and at least one non-missing post-baseline were included in analysis.
Measure: Number; unit: participants
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 357 | 177
participants | 69 | 31
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.639, Fisher Exact

12. Secondary Outcome: Rate of Total Symptomatic and Nocturnal Hypoglycemia Events (Adjusted by 1 Year)
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 mmol/L). The overall yearly rates (events/participant/year) of those hypoglycemic events, calculated as, for each participant, the number of episodes times 365.25 and then divided by the participants treatment duration, will be summarized, and analyzed by a negative-binomial regression model with treatment as fixed effects and log of (participant's treatment duration/365.25) as an offset variable. A nocturnal hypoglycemic event is defined as any total hypoglycemia event that occurred between bedtime and waking.
Time Frame: Baseline through 24 weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and at least one non-missing post-baseline hypoglycemic event.
Measure: Least Squares Mean (Standard Error); unit: events/participant/year
Arm/Group | LY2963016 | Lantus®
Number analyzed (Participants) | 359 | 177
events/participant/year
  Total hypoglycemia | 1.37 (0.228) | 1.15 (0.280)
  Nocturnal Hypoglycemia | 0.47 (0.132) | 0.39 (0.110)
Statistical Analysis 1: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.143, Wilcoxon (Mann-Whitney); Relative Ratio = 1.19, 95% CI 2-sided [0.74 to 1.92]
Statistical Analysis 2: Comparison: LY2963016 vs Lantus®; Test type: Superiority; p = 0.945, Wilcoxon (Mann-Whitney); Relative Ratio = 1.22, 95% CI 2-sided [0.67 to 2.23]

ADVERSE EVENTS:
Time Frame: Baseline Up To 28 Weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | LY2963016 | Lantus®
All-Cause Mortality (participants affected / at risk) | 0/359 | 0/177
Serious Adverse Events (participants affected / at risk) | 28/359 | 14/177
Other Adverse Events (participants affected / at risk) | 194/359 | 95/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 (N=359) | Lantus® (N=177)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Malignant glaucoma (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 5 (6) | 2 (2)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2963016 (N=359) | Lantus® (N=177)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (3) | 2 (3)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 4 (4) | 1 (2)
Cataract (Eye disorders) | 5 (6) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 10 (14) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (8) | 3 (3)
Toothache (Gastrointestinal disorders) | 9 (11) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 3 (3)
Chest pain (General disorders) | 7 (7) | 2 (2)
Hunger (General disorders) | 2 (3) | 2 (2)
Injection site pain (General disorders) | 15 (19) | 5 (5)
Injection site pruritus (General disorders) | 4 (5) | 1 (1)
Injection site rash (General disorders) | 4 (7) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 6 (6)
Gastroenteritis (Infections and infestations) | 4 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8) | 7 (7)
Otitis media (Infections and infestations) | 1 (1) | 2 (2)
Periodontitis (Infections and infestations) | 3 (4) | 4 (5)
Pharyngitis (Infections and infestations) | 9 (9) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 3 (4)
Pulpitis dental (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 5 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 73 (80) | 32 (38)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Vaginal infection (Infections and infestations) | 1/150 (1) | 1/79 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Blood pressure increased (Investigations) | 4 (4) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 14 (14) | 11 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (5)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 2 (3)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 8 (10) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal cyst (Renal and urinary disorders) | 3 (3) | 4 (4)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 2 (2)
Balanoposthitis (Reproductive system and breast disorders) | 0/209 (0) | 1/98 (1)
Prostatic calcification (Reproductive system and breast disorders) | 0/209 (0) | 1/98 (1)
Uterine atrophy (Reproductive system and breast disorders) | 0/150 (0) | 1/79 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 2 (2)
Arteriosclerosis (Vascular disorders) | 3 (3) | 2 (3)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 20 (20) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03338010/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT03338010/SAP_001.pdf